CLINICAL TRIAL: NCT05880836
Title: In Line Aerosol Nebulization With High Flow
Acronym: ILAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Aerogen (Industry)
Responsible Party: Principal Investigator, Igor Barjaktarevic, MD, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-001966
Record Dates: First submitted 2023-03-08; First posted 2023-05-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-03

CONDITIONS: Hypoxemic Respiratory Failure; Airway Obstruction
MeSH Terms: conditions — Respiratory Insufficiency; Airway Obstruction

STUDY DESIGN:
Intervention Model Description: HFNC with trans-nasal aerosol delivery is a multi-center trial comparing nebulization of medications via trans-nasal delivery with vibrating mesh nebulizer to standard jet nebulization in patients with mild or moderate hypoxemic respiratory failure (with or without acute hypercapnic respiratory failure) treated with HFNC. The crossover nature of the study is reflected in the universal application of bronchodilators via both study interventions (HFNC/VMN and FM/SJN) in all subjects but in variable order depending on the randomization of subjects into Path A or Path B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Path A (vibrating mesh nebulizer (VMN) with the high flow nasal cannula) (Experimental): Enrolled patients will receive two standard forms of inhaled medications as ordered by the physician. Patients will be randomized into two paths of the cross over study. There will be no blinding involved in this randomization. Path A will have medications delivered trans-nasally in line via the vibrating mesh nebulizer (VMN) with the high flow nasal cannula followed by standard jet nebulization (SJN) with face mask at the next time of medication dosing 3-6 hours later.
  Interventions: Device: nebulizer via in-line drug delivery maintaining high-flow nasal cannula oxygen; Device: standard jet nebulization (SJN) with face mask
- Path B (standard jet nebulization (SJN) with face mask) (Active Comparator): Path B will receive standard jet nebulization without HFNC followed by the trans-nasal in line nebulization via the HFNC. Patients agreed to enroll in day 2 of the trial will have their clinical path alternated in attempt to control for diurnal variability. All patients will also receive as-needed nebulized treatments as well as usual supportive care provided by respiratory therapists. As needed therapy will be delivered via the method of the current arm of the study they are in, and the washout period will subsequently reset.
  Interventions: Device: nebulizer via in-line drug delivery maintaining high-flow nasal cannula oxygen; Device: standard jet nebulization (SJN) with face mask

INTERVENTIONS:
Device: nebulizer via in-line drug delivery maintaining high-flow nasal cannula oxygen — nebulized delivery of bronchodilator via in-line drug delivery maintaining high-flow nasal cannula oxygen
Device: standard jet nebulization (SJN) with face mask — standard jet nebulization delivery of bronchodilator

SUMMARY:
The objective of ILAN is to assess the safety, feasibility and bronchodilator efficacy of in-line bronchodilator nebulizer delivery with VMN via HFNC system in hypoxemic respiratory failure patients treated with bronchodilators and compare this method to standard-nebulization using a jet nebulizer with a facial mask. The investigators hypothesized that aerosol nebulization using HFNC/VMN represents safer and more convenient approach in hypoxemic respiratory failure patients in comparison to conventional therapy while providing similar bronchodilator efficacy.

DETAILED DESCRIPTION:
Objective: To evaluate the safety and feasibility of a novel approach to nebulization treatment via the nasal route in patients with severe hypoxemic respiratory failure dependent on high flow oxygen.

Hypothesis: In-line vibrating mesh nebulizer delivery via HFNC systems is a safe, feasible and efficacious approach in comparison to traditional jet nebulizer delivered nebulization in hypoxemic respiratory failure patients whose usual care includes nebulized drugs.

Specific Aims:

1. To evaluate the safety and feasibility of administering vibrating mesh nebulizer-delivered therapy in patients with acute hypoxemic respiratory failure requiring high flow nasal cannula.
2. To evaluate the effect of trans-nasal nebulization on patient comfort and satisfaction with therapy in comparison with standard jet nebulization.
3. To evaluate differences in resource utilization between patients receiving standard jet nebulization and ILAN with HF, including time spent at the bedside by the respiratory therapist (RT) for delivery of the medication and any additional time gathering setting up and cleaning.
4. To evaluate patient and therapist perceptions and preference on the various delivery methods of aerosol delivery.

Study Design: ILAN is a double-crossover, multi-center trial evaluating the safety and feasibility of in line nebulized medication with high flow nasal canula in comparison to standard jet nebulizer therapy in acute respiratory failure requiring the utilization of high flow nasal cannula.

Intervention: Enrolled patients will receive two standard forms of inhaled medications as ordered by the physician. Patients will be randomized into two paths of the cross over study. There will be no blinding involved in this randomization. Path A will have medications delivered trans-nasally in line via the vibrating mesh nebulizer (VMN) with the high flow nasal cannula followed by standard jet nebulization (SJN) with face mask at the next time of medication dosing 3-6 hours later. Path B will receive standard jet nebulization without HFNC followed by the trans-nasal in line nebulization via the HFNC. Patients selected to enroll in day 2 of the trial will have their clinical path alternated in attempt to control for diurnal variability. All patients will also receive as-needed nebulized treatments as well as usual supportive care provided by respiratory therapists. As needed therapy will be delivered via the method of the current arm of the study they are in, and the washout period will subsequently reset.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patients with mild or moderate hypoxemic respiratory failure (with or without acute hypercapnic respiratory failure) treated with HFNC.
* Nebulizer therapy ordered by the primary team with at least one dose delivered prior to the enrollment into the study
* Patients must be on ordered nebulized albuterol, levalbuterol, ipratropium or ipratropium/albuterol combination with a maximum of Q3 or a minimum of Q6 hour frequencies.
* For Respiratory Therapists: They must be employees of SMICU or RRMC.

Exclusion Criteria:

* Lack of hypoxemia defined as SpO2> 92% on room air
* Severe hypoxemia defined by PaO2/FiO2<100 or SpO2<92% on HFNC settings: ≥ FiO2 80% or higher and O2 flow 40L/min
* HFNC O2 delivery via tracheostomy
* COVID-19 positive status (within 3 weeks prior to the enrollment)
* Respiratory distress, defined by respiratory rate > 24 breath per minute
* Hemodynamic instability defined by the use of two or more vasopressor medications
* Presence of nasal obstruction that may pose a risk for inadequate nebulizer delivery in the opinion of the investigator
* Pulmonary comorbidities that, in the opinion of the investigator or clinical team, can pose a risk to subject safety or interfere with the subject's ability to complete the study procedures.
* Moribund patient not expected to survive >24 hours
* Inability to obtain informed consent from patient
* Respiratory therapists who are unwilling to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Maximal decrease in SpO2 during nebulization with jet nebulizer vs. inline via HFNC compared to the baseline SpO2 values prior to the nebulization therapy | up to 48 hours
  Primary Outcome

SECONDARY OUTCOMES:
Proportion of patients with documented hypoxemia (<88%) during the nebulization | up to 48 hours
  Safety Outcome
Duration of hypoxemic episodes with SpO2<88% during the nebulization delivery | up to 48 hours
  Safety Outcome
Lowest absolute desaturation from the beginning until completion of nebulizer treatment compared to the baseline SpO2 values defined as the lowest adequately measured SpO2 within two minutes prior to the nebulization | up to 48 hours
  Safety Outcome
Increase in respiratory rate from the baseline during the nebulization by >10% | up to 48 hours
  Safety Outcome
Change in respiratory rate during nebulization compared to the baseline rate | up to 48 hours
  Safety Outcome
Requirement for additional interventions to maintain patient's safety during the nebulization | up to 48 hours
  Safety Outcome: (Increased O2 flow (yes/know and rate increase) or increased O2 FiO2 (yes/know and rate increase) )
Need to increase O2 support after the nebulization therapy to maintain SpO2>88% | up to 48 hours
  Safety Outcome
Nosebleed within 2 hours of nebulizer delivery | up to 48 hours
  Safety Outcome
ROX score | up to 48 hours
  Safety Outcome (While not externally validated, the ROX Index is a simple bedside calculation using three clinical variables and is one easy way to summarize a patient's degree of hypoxemic respiratory failure - gives risk of intubation - low to high)

OTHER OUTCOMES:
Portion of patients able to complete the nebulization therapy | up to 48 hours
  Feasibility Outcome
Patient satisfactory survey score | up to 48 hours
  Feasibility Outcome: (5 question, 7-point scale ranging from very uncomfortable to very comfortable)
Modified BORG score | up to 48 hours
  Safety Outcome (Introduced by Gunnar Borg, rates exertion on a scale of 6-20, from lowest to highest)
Compliance with the study protocol | up to 48 hours
  Feasibility Outcome (number of study drug doses which are missed during the study period)
Duration of nebulizer delivery | up to 48 hours
  Feasibility Outcome
Respiratory therapist time utilization as reflected in the total time spent delivering the nebulization in 2-minute increments | up to 48 hours
  Feasibility Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Igor Barjaktarevic, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan Medical Center at UCLA, Los Angeles, California
  - Santa Monica UCLA, Santa Monica, California

IPD SHARING:
Plan to Share IPD: Yes
as below
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the study completion, for 3 years
Access Criteria: direct contact with the study team

REFERENCES:
- [Background] 1. Rochwerg, B. Intensive Care Med, 2020 2. Li, J. Respir Care, 2021 3. Reminiac, F. Ann Intensive Care, 2018 4. Li, J. Crit Care, 2020. 5. Dugernier, J., J Aerosol Med Pulm Drug Deliv, 2019 6. Leung, C.C.H. J Hosp Infect, 2019 7. Reminiac, F., J Aerosol Med Pulm Drug Deliv, 2016 8. Berlinski, A. Respir Care, 2013 9. Ari, A., J Aerosol Med Pulm Drug Deliv, 2015 10. Ari, A., Respir Care, 2010 11. Alcoforado, L., Pharmaceutics, 2019 12. Bennett, G., Intensive Care Med Exp, 2019 13. Dugernier, J.,J Aerosol Med Pulm Drug Deliv, 2017 14. Zielinski, J., Chest, 1995 15. Ringbaek, T. and K. Viskum, Respir Med, 2003 16. Rezaie, N. J Res Med Sci, 2013 17. Rennard, S.I., Chest, 1996 18. Ogale, S.S., Chest, 2010 19. Drake, M.G., Ann Am Thorac Soc, 2018 20. Valencia-Ramos, J., Respir Care, 2018